CLINICAL TRIAL: NCT05517746
Title: Randomized, Placebo-controlled, Double-blind Study to Investigate the Safety, Tolerability and Pharmacokinetics of Increasing Single and Multiple Oral Doses of BAY 2395840 Including the Relative Bioavailability Between Solution and Tablet Formulation and the Effect of Food on the Pharmacokinetics of BAY 2395840 in Healthy Men
Brief Title: Study on the Safety of the Drug BAY2395840 at Different Doses, the Way the Body Absorbs, Distributes and Excretes the Drug Including the Effect of Its Formulation (Tablet or Liquid) and the Effect of Food on the Absorption, Distribution or Excretion of the Drug in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 19634; 2019-002573-65 (EudraCT Number)
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Group 1 (Experimental): Participants received BAY2395840 dose A as tablets under diet 1 conditions (Period 1). After the safety assessment for Period 1 and a washout period of at least 14 days participants were re-dosed with the same BAY2395840 dose A1 as oral solution under diet 1 conditions (Period 2)
  Interventions: Drug: BAY2395840 tablet; Drug: BAY2395840 oral solution
- Group 2 (Experimental): Participants received BAY2395840 dose C as tablets under diet 1 conditions.
  Interventions: Drug: BAY2395840 tablet
- Group 3 (Experimental): Participants received BAY2395840 dose E as tablets under diet 1 conditions.
  Interventions: Drug: BAY2395840 tablet
- Group 4 (Experimental): Participants received BAY2395840 dose H as tablets under diet 1 conditions
  Interventions: Drug: BAY2395840 tablet
- Group 5 (Experimental): Participants received BAY2395840 dose B as tablets on Day 1 after diet 2, on Days 2 to 7 under diet 1 conditions
  Interventions: Drug: BAY2395840 tablet
- Group 6 (Experimental): Participants received BAY2395840 dose C as tablets on Day 1 after diet 2, on Days 2 to 7 under diet 1 conditions
  Interventions: Drug: BAY2395840 tablet
- Group 7 (Experimental): Participants received BAY2395840 dose I as tablets under diet 1 conditions
  Interventions: Drug: BAY2395840 tablet
- Group 8 (Experimental): Participants received BAY2395840 dose G as tablets on Day 1, followed by 3 BAY395840 doses of dose F as tablets on Days 2 to 4 and subsequently 7 further BAY395840 doses of dose G as tablets on Days 5 to 11 under diet 1 conditions
  Interventions: Drug: BAY2395840 tablet
- Placebo matching Group 1 (Placebo Comparator): Participants received a dose of placebo as tablets under diet 1 conditions (Period 1). After the safety assessment for Period 1 and a washout period of at least 14 days participants were re-dosed with a single dose of placebo as oral solution under under diet 1 conditions (Period 2)
  Interventions: Drug: Placebo oral solution; Drug: Placebo tablet
- Placebo matching Group 2 to 4 and Group 7 (Placebo Comparator): Participants received a dose of Placebo as tablets under diet 1 conditions
  Interventions: Drug: Placebo tablet
- Placebo matching Group 5 and 6 (Placebo Comparator): Participants received Placebo as tablets on Day 1 after diet 2, on Days 2 to 7 under diet 1 conditions
  Interventions: Drug: Placebo tablet
- Placebo matching Group 8 (Placebo Comparator): Participants received a dose of Placebo as tablets on Day 1, followed by 3 doses of Placebo as tablets on Days 2 to 4 and subsequently 7 further doses of Placebo as tablets on Days 5 to 11 under diet 1 conditions.
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: BAY2395840 tablet — tablets, oral administration
  Arms: Group 1; Group 2; Group 3; Group 4; Group 5; Group 6; Group 7; Group 8
Drug: BAY2395840 oral solution — solution, oral administration
  Arms: Group 1
Drug: Placebo oral solution — Placebo matching BAY2395840, oral administration
  Arms: Placebo matching Group 1
Drug: Placebo tablet — Placebo matching BAY2395840, oral administration
  Arms: Placebo matching Group 1; Placebo matching Group 2 to 4 and Group 7; Placebo matching Group 5 and 6; Placebo matching Group 8

SUMMARY:
Researchers are looking for a better way to treat people who have endometriosis, a condition in which tissue similar to the lining of the uterus starts to grow in places outside of the uterus. The study treatment, BAY2395840, is being developed to help block certain proteins from causing inflammation and pain in people with endometriosis. But, this is the first time that researchers will study BAY2395840 in humans.

In this study, the researchers will learn how safe BAY2395840 is for the participants to take. They will also learn what happens to BAY2395840 in the body. The study will include about 56 healthy adult men.

All of the participants will take increasing doses of BAY2395840, or a placebo. A placebo looks like a treatment but does not have any medicine in it. Some of the participants will take their study treatment 1 time under diet 1 conditions. The other participants will take their study treatment 7 times with diet 1 or diet 2.

The participants will take BAY2395840 or the placebo as tablets or as a liquid by mouth. The participants will stay at the study site for up to 11 days . After that, they will visit the study site 1 more time. Each participant will be in the study for up to about 14 weeks.

During the study, the doctors will collect blood and urine samples and check the participants' overall health and heart health. The participants will answer questions about how they are feeling, what medications they are taking, and what adverse events they are having. An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Male participants of age 18 to 45 years (inclusive), at the time of signing the informed consent.
* Body mass index (BMI) ≥18 kg/m^2 and ≤30 kg/m^2.
* Participants who are overtly healthy.
* Race: White.
* Male participants of reproductive potential who are sexually active must agree to use contraception methods.

Exclusion Criteria:

* Any findings from the medical examination (including medical history, physical examination, vital signs, laboratory tests and ECG) deviating from normal and deemed to be of clinical relevance by the investigator.
* Any known disease that was forbidden in the study as specified in study protocol.
* Any medication or drug use that was forbidden in the study as specified in study protocol.
* Any abnormal finding in Electrocardiogram (ECG), blood pressure or heart rate.
* Any clinical relevant deviation from normal range of laboratory parameters at screening.
* History of COVID-19.
* Prior contact with SARS-CoV-2 positive person or COVID-19 patient within the last 4 weeks prior admission to the ward.
* Positive SARS-CoV-2 viral RNA test.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events | Up to 14 days after end of treatment with study medication in the respective period.
Number of participants with treatment-emergent adverse events, categorized by severity. | Up to 14 days after end of treatment with study medication in the respective period.

SECONDARY OUTCOMES:
Maximum observed drug concentration in plasma (Cmax) after single dose of BAY2395840 | Predose up to 192 hours
Area under the concentration vs. time curve from zero to infinity (AUC) in plasma after single dose of BAY2395840 | Predose up to 192 hours
Area under the plasma concentration-time curve from zero to 24 hours AUC (0-24) after single dose of BAY2395840 | Pre-dose and up to 24 hours post dose
  AUC from time 0 to 24 hours
Maximum observed drug concentration in plasma (Cmax) after multiple doses of BAY2395840 | Predose up to 192 hours
Area under the plasma concentration-time curve over the last 24-h dosing interval AUC(0-24)in plasma after multiple doses of BAY2395840 | Pre-dose and up to 24 hours post dose
  AUC from time 0 to 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.